CLINICAL TRIAL: NCT02266706
Title: A Phase 1, Non-comparative, Open-label Study to Characterize the Pharmacokinetics of a Single Intravenous Dose of Ceftolozane/Tazobactam in Pediatric Patients Receiving Standard of Care Antibiotic Therapy for Proven or Suspected Gram-negative Infection or for Peri-operative Prophylaxis
Brief Title: Pharmacokinetic and Safety Study of Ceftolozane/Tazobactam in Pediatric Participants Receiving Antibiotic Therapy for Proven or Suspected Gram-negative Infection or for Peri-operative Prophylaxis (MK-7625A-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7625A-010; CXA-PEDS-13-08 (Other: Cubist Pharmaceuticals LLC Protocol Number); 2014-003485-24 (EudraCT Number); MK-7625A-010 (Other: Merck Protocol Number); NCT02725216 (obsolete NCT alias)
Record Dates: First submitted 2014-09-22; First posted 2014-10-17 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Proven or Suspected Gram-negative Bacterial Infection; Peri-operative Prophylaxis
MeSH Terms: interventions — ceftolozane; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: ≥12 to <18 years TOL/TAZ 1000/500 mg FDC (Experimental): Participants ≥12 to <18 years of age received a single dose of ceftolozane/tazobactam (TOL/TAZ) 1000/500 mg FDC as a 60-minute infusion on Day 1.
  Interventions: Drug: Ceftolozane/Tazobactam 1000/500 mg
- Cohort 2: ≥7 to <12 years TOL/TAZ 18/9 mg/kg (Experimental): Participants ≥7 to <12 years of age received a single dose of TOL/TAZ 18/9 mg/kg as a 60-minute infusion on Day 1.
  Interventions: Drug: Ceftolozane/Tazobactam 18/9 mg/kg
- Cohort 3: ≥2 to <7 years TOL/TAZ 18/9 or 30/15 mg/kg (Experimental): Participants ≥2 to <7 years of age received a single dose of TOL/TAZ 18/9 mg/kg as a 60-minute infusion on Day 1. Participants in this cohort enrolled after interim analysis for Cohort 3 received TOL/TAZ 30/15 mg/kg.
  Interventions: Drug: Ceftolozane/Tazobactam 30/15 mg/kg; Drug: Ceftolozane/Tazobactam 18/9 mg/kg
- Cohort 4: ≥3 months to <2 years TOL/TAZ 18/9 or 30/15 mg/kg (Experimental): Participants ≥3 months to <2 years of age received a single dose of TOL/TAZ 18/9 mg/kg as a 60-minute infusion on Day 1. Participants in this cohort enrolled after interim analysis for Cohort 3 received TOL/TAZ 30/15 mg/kg.
  Interventions: Drug: Ceftolozane/Tazobactam 30/15 mg/kg; Drug: Ceftolozane/Tazobactam 18/9 mg/kg
- Cohort 5: birth to <3 months TOL/TAZ 20/10 mg/kg (Experimental): Participants from birth (>32 weeks gestation, 7 days postnatal) to <3 months of age received a single dose of TOL/TAZ 20/10 mg/kg as a 60-minute infusion on Day 1. After interim analysis for Cohort 4, the original regimen of TOL/TAZ 12/6 mg/kg was changed to TOL/TAZ 20/10.
  Interventions: Drug: Ceftolozane/Tazobactam 20/10 mg/kg
- Cohort 6: birth to <3 months TOL/TAZ 12/6 or 20/10 mg/kg (Experimental): Participants from birth (≤32 weeks gestation, 7 days postnatal) to <3 months of age with creatinine clearance =20 - 49 mL/min/1.73 m^2 received a single dose of TOL/TAZ 12/6 mg/kg as a 60-minute infusion on Day 1; participants with creatinine clearance ≥50 mL/min/1.73 m^2 received a single dose of TOL/TAZ 20/10 mg/kg as a 60-minute infusion on Day 1. After interim analysis for Cohort 4, the original regimen of TOL/TAZ 12/6 was changed to TOL/TAZ 20/10 mg/kg for participants with creatinine clearance ≥50 mL/min/1.73 m^2.
  Interventions: Drug: Ceftolozane/Tazobactam 20/10 mg/kg; Drug: Ceftolozane/Tazobactam 12/6 mg/kg

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam 1000/500 mg — A fixed dose combination (FDC) of 1000 mg ceftolozane and 500 mg tazobactam as a 60 minute infusion.
  Arms: Cohort 1: ≥12 to <18 years TOL/TAZ 1000/500 mg FDC
Drug: Ceftolozane/Tazobactam 30/15 mg/kg — A FDC of 30 mg/kg of ceftolozane and 15 mg/kg of tazobactam as a 60 minute infusion.
  Arms: Cohort 3: ≥2 to <7 years TOL/TAZ 18/9 or 30/15 mg/kg; Cohort 4: ≥3 months to <2 years TOL/TAZ 18/9 or 30/15 mg/kg
Drug: Ceftolozane/Tazobactam 20/10 mg/kg — A FDC of 20 mg/kg of ceftolozane and 10 mg/kg of tazobactam as a 60 minute infusion.
  Arms: Cohort 5: birth to <3 months TOL/TAZ 20/10 mg/kg; Cohort 6: birth to <3 months TOL/TAZ 12/6 or 20/10 mg/kg
Drug: Ceftolozane/Tazobactam 18/9 mg/kg — A FDC of 18 mg/kg of ceftolozane and 9 mg/kg of tazobactam as a 60 minute infusion.
  Arms: Cohort 2: ≥7 to <12 years TOL/TAZ 18/9 mg/kg; Cohort 3: ≥2 to <7 years TOL/TAZ 18/9 or 30/15 mg/kg; Cohort 4: ≥3 months to <2 years TOL/TAZ 18/9 or 30/15 mg/kg
Drug: Ceftolozane/Tazobactam 12/6 mg/kg — A FDC of 12 mg/kg of ceftolozane and 6 mg/kg of tazobactam as a 60 minute infusion.
  Arms: Cohort 6: birth to <3 months TOL/TAZ 12/6 or 20/10 mg/kg

SUMMARY:
The purpose of this study was to assess the pharmacokinetics, safety, and tolerability of a single intravenous dose of ceftolozane/tazobactam (MK-7625A) in pediatric participants. In each of the 6 age cohorts, an interim analysis of pharmacokinetics (PK) and safety data was conducted after approximately 3 participants had received the initially proposed dose. The interim analysis was to determine whether the initial dose was appropriate based on pre-defined criteria. If data from the interim analysis demonstrated that the initially proposed dose met the above criteria, enrollment was to continue with the same dose administered to approximately 3 additional participants of the same age range. However, if the interim analysis demonstrated that a new optimized dose was required, the new dose was to be administered to approximately 3 additional participants of the same age range.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or non-pregnant females from birth to <18 years of age
2. Receiving standard of care antibiotic therapy for suspected or diagnosed Gram-negative infection or for peri-operative prophylaxis
3. Groups 1-4: Calculated creatinine clearance rate (CLCR) ≥ 80 ml/min/1.73m2 at baseline
4. Group 5: CLCR ≥ 50 ml/min/1.73m2 at baseline
5. Group 6: CLCR ≥ 20 ml/min/1.73m2 at baseline

Key Exclusion Criteria:

1. Known allergy/hypersensitivity to any β-lactam antibacterial
2. History of clinically significant renal, hepatic, or hemodynamic instability
3. Planned use of cardiopulmonary bypass or dialysis
4. Planned blood transfusion within 24 hours of study drug administration
5. Clinically significant abnormal laboratory test results not related to the underlying infection
6. Receipt of piperacillin/tazobactam within 24 hours of study drug administration
7. Likely to be at risk of hemodynamic disturbance following collection of the required PK blood samples

Ages: 7 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Bradley JS, Ang JY, Arrieta AC, Larson KB, Rizk ML, Caro L, Yang S, Yu B, Johnson MG, Rhee EG. Pharmacokinetics and Safety of Single Intravenous Doses of Ceftolozane/Tazobactam in Children With Proven or Suspected Gram-Negative Infection. Pediatr Infect Dis J. 2018 Nov;37(11):1130-1136. doi: 10.1097/INF.0000000000002170. PMID 30153232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for eligibility within 48 hours prior to study drug administration.
Pre-assignment Details: After interim analysis, dose level adjustments were made to some groups based on safety and pharmacokinetics targets. Thus, the initial 6 cohorts were expanded to a total of 9 cohorts for analysis.
Groups:
- Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg: Participants ≥7 to <12 years of age received a single dose of ceftolozane/tazobactam 18/9 mg/kg as a 60-minute infusion on Day 1.
- Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg: Participants ≥2 to <7 years of age received a single dose of ceftolozane/tazobactam 18/9 mg/kg as a 60-minute infusion on Day 1.
- Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg: Participants ≥2 to <7 years of age received a single dose of ceftolozane/tazobactam 30/15 mg/kg as a 60-minute infusion on Day 1.
- Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg: Participants ≥3 months to <2 years of age received a single dose of ceftolozane/tazobactam 18/9 mg/kg as a 60-minute infusion on Day 1.
- Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg: Participants ≥3 months to <2 years of age received a single dose of ceftolozane/tazobactam 30/15 mg/kg as a 60-minute infusion on Day 1.
- Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg: Participants from birth (>32 weeks gestation, 7 days postnatal) to <3 months of age received a single dose of ceftolozane/tazobactam 20/10 mg/kg as a 60-minute infusion on Day 1.
- Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg: Participants from birth (≤32 weeks gestation, 7 days postnatal) to <3 months of age with creatinine clearance of 20 - 49 mL/min/1.73 m^2 received a single dose of ceftolozane/tazobactam 12/6 mg/kg as a 60-minute infusion on Day 1.
- Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg: Participants from birth (≤32 weeks gestation, 7 days postnatal) to <3 months of age with creatinine clearance ≥50 mL/min/1.73 m^2 received a single dose of ceftolozane/tazobactam 20/10 mg/kg as a 60-minute infusion on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Started | 6 | 7 | 4 | 4 | 1 | 7 | 8 | 2 | 4
Treated | 6 | 6 | 3 | 3 | 1 | 5 | 7 | 2 | 4
Completed | 6 | 6 | 3 | 3 | 1 | 5 | 7 | 2 | 4
Not Completed | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Screen failure | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Enrollment in another study | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Total
Number analyzed (Participants) | 6 | 7 | 4 | 4 | 1 | 7 | 8 | 2 | 4 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.1 (1.4) | 8.5 (1.2) | 5.5 (0.8) | 4.8 (1.8) | 0.9 (0.0) | 0.9 (0.7) | 0.1 (0.0) | 0.1 (0.0) | 0.2 (0.1) | 4.8 (5.6)
Age, Customized [Count of Participants; unit: Participants]
  Newborns (0-27days) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 1 | 6 | 6 | 2 | 4 | 19
  Children (2-11 years) | 0 | 7 | 4 | 4 | 0 | 1 | 0 | 0 | 0 | 16
  Adolescents (12-17 years) | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 3 | 0 | 2 | 4 | 0 | 3 | 22
  Male | 1 | 4 | 2 | 1 | 1 | 5 | 4 | 2 | 1 | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 8
  White | 5 | 7 | 4 | 2 | 0 | 6 | 7 | 0 | 0 | 31
  Other | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Ceftolozane
Description: Blood was collected for the determination of Cmax of ceftolozane. Cmax is expressed as geometric least-squares mean and confidence interval based on back-transformed least-squares mean and confidence interval from linear mixed-effects model with group fixed effect performed on natural log-transformed values.
Time Frame: Predose and 0.5, 1, 2, 4, and 6 hours after the start of infusion for Cohorts 1 to 4 and 1, 2, and 6 hours after start of infusion for Cohorts 5 and 6.
Population: The pharmacokinetics population included enrolled participants who received a full dose of study drug and had blood samples with quantifiable plasma levels at Cmax and at least 2 time points after Cmax, and were evaluable for the outcome measure.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
μg/mL | 63.5 [50.2 to 80.4] | 56.2 [45.3 to 69.7] | 51.4 [37.9 to 69.7] | 96.6 [71.2 to 131] | 50.5 [29.8 to 85.6] | 91.3 [72.1 to 116] | 45.0 [36.3 to 55.9] | 34.9 [24.1 to 50.7] | 45.2 [33.3 to 61.2]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Tazobactam
Description: Blood was collected for the determination of Cmax of tazobactam. Cmax is expressed as geometric least-squares mean and confidence interval based on back-transformed least-squares mean and confidence interval from linear mixed-effects model with group fixed effect performed on natural log-transformed values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
μg/mL | 14.0 [8.59 to 22.9] | 9.25 [5.92 to 14.5] | 15.7 [8.36 to 29.6] | 24.8 [13.2 to 46.6] | 11.6 [3.88 to 34.7] | 22.4 [13.8 to 36.6] | 11.7 [7.48 to 18.3] | 6.87 [3.17 to 14.9] | 12.1 [6.43 to 22.7]

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Ceftolozane
Description: Blood was collected for the determination of Tmax of ceftolozane.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours | 1.02 [1.00 to 1.10] | 1.07 [0.58 to 1.13] | 1.02 [1.02 to 1.03] | 1.03 [1.03 to 1.12] | 1.00 [1.00 to 1.00] | 1.05 [0.58 to 1.95] | 1.08 [0.95 to 1.90] | 1.80 [1.03 to 2.57] | 1.07 [1.07 to 1.18]

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Tazobactam
Description: Blood was collected for the determination of Tmax of tazobactam.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours | 1.00 [0.50 to 1.10] | 1.07 [0.58 to 1.13] | 1.02 [1.02 to 1.03] | 1.03 [1.03 to 1.12] | 1.00 [1.00 to 1.00] | 1.05 [0.58 to 1.95] | 1.08 [0.95 to 1.33] | 3.89 [1.03 to 6.75] | 1.07 [1.07 to 1.18]

5. Primary Outcome: Plasma Concentration at the Last Quantifiable Concentration (Clast) of Ceftolozane
Description: Blood was collected for the determination of Clast of ceftolozane. Clast is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
μg/mL | 4.01 (40.4) | 2.85 (37.3) | 2.47 (29.1) | 5.69 (59.5) | 2.53 (NA) — Cannot be calculated for n=1 | 5.72 (96.1) | 8.70 (49.1) | 10.2 (49.2) | 6.26 (39.2)

6. Primary Outcome: Plasma Concentration at the Last Quantifiable Concentration (Clast) of Tazobactam
Description: Blood was collected for the determination of Clast of tazobactam. Clast is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
μg/mL | 0.232 (52.2) | 0.420 (188.6) | 0.137 (24.1) | 0.327 (62.7) | 0.224 (NA) — Cannot be calculated for n=1 | 0.401 (90.5) | 0.657 (169.2) | 3.66 (57.6) | 0.266 (81.3)

7. Primary Outcome: Time of Last Sampling Point (Tlast) of Ceftolozane
Description: Blood was collected for the determination of Tlast of ceftolozane.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours | 6.00 [5.85 to 6.03] | 6.01 [5.82 to 6.15] | 6.08 [5.85 to 6.25] | 5.77 [5.72 to 5.93] | 6.00 [6.00 to 6.00] | 6.00 [5.72 to 6.75] | 6.01 [5.88 to 6.18] | 6.40 [6.05 to 6.75] | 5.85 [5.72 to 6.02]

8. Primary Outcome: Time of Last Sampling Point (Tlast) of Tazobactam
Description: Blood was collected for the determination of Tlast of tazobactam.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours | 4.15 [4.00 to 6.00] | 3.10 [2.02 to 4.15] | 5.85 [4.03 to 6.08] | 5.72 [3.85 to 5.93] | 4.00 [4.00 to 4.00] | 5.02 [4.02 to 5.75] | 5.95 [2.18 to 6.10] | 6.40 [6.05 to 6.75] | 5.85 [5.72 to 6.02]

9. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUClast) of Ceftolozane
Description: Blood was collected for the determination of AUC from time zero to the last quantifiable concentration of ceftolozane. AUC0-last is expressed as geometric least squares mean and confidence interval based on back-transformed least-squares mean and confidence interval from linear mixed-effects model with group fixed effect performed on natural log-transformed values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Hours*μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours*μg/mL | 124 [103 to 150] | 102 [86.2 to 121] | 94.2 [74.1 to 120] | 172 [135 to 219] | 98.8 [65.1 to 150] | 178 [148 to 214] | 131 [111 to 155] | 118 [88.2 to 159] | 119 [93.7 to 151]

10. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUClast) of Tazobactam
Description: Blood was collected for the determination of AUC from time zero to the last quantifiable concentration of tazobactam. AUC0-last is expressed as geometric least squares mean and confidence interval based on back-transformed least-squares mean and confidence interval from linear mixed-effects model with group fixed effect performed on natural log-transformed values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Hours*μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours*μg/mL | 17.3 [10.7 to 27.9] | 9.69 [6.27 to 15.0] | 17.6 [9.53 to 32.7] | 28.5 [15.4 to 52.8] | 14.8 [5.08 to 42.9] | 28.9 [18.0 to 46.6] | 21.3 [13.8 to 33.0] | 21.6 [10.2 to 45.9] | 21.9 [11.8 to 40.6]

11. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC0-inf) of Ceftolozane
Description: Blood was collected for the determination of AUC from time zero extrapolated to infinity of ceftolozane. AUC0-inf is expressed as geometric least squares mean and confidence interval based on back-transformed least-squares mean and confidence interval from linear mixed-effects model with group fixed effect performed on natural log-transformed values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Hours*μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours*μg/mL | 133 [104 to 171] | 107 [85.7 to 135] | 99.4 [72.2 to 137] | 186 [135 to 255] | 103 [59.4 to 180] | 202 [158 to 259] | 164 [131 to 205] | 165 [112 to 244] | 137 [99.6 to 189]

12. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC0-inf) of Tazobactam
Description: Blood was collected for the determination of AUC from time zero extrapolated to infinity of tazobactam. AUC0-inf is expressed as geometric least squares mean and confidence interval based on back-transformed least-squares mean and confidence interval from linear mixed-effects model with group fixed effect performed on natural log-transformed values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Hours*μg/mL
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 1 | 5 | 5 | 1 | 3
Hours*μg/mL | 17.5 [12.6 to 24.2] | 10.2 [6.68 to 15.5] | 17.8 [11.7 to 27.0] | 28.9 [19.0 to 43.9] | 14.9 [7.21 to 30.9] | 29.9 [21.6 to 41.4] | 24.9 [18.0 to 34.4] | 77.6 [37.5 to 161] | 22.3 [14.7 to 34.0]

13. Primary Outcome: Elimination Half-life (t1/2) of Ceftolozane
Description: Blood was collected for the determination of t1/2 of ceftolozane. t1/2 is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
Hours | 1.45 (16.7) | 1.29 (9.6) | 1.34 (14.0) | 1.48 (35.5) | 1.30 (NA) — Cannot be calculated for n=1 | 1.63 (69.0) | 2.21 (37.6) | 3.14 (0.9) | 1.73 (29.7)

14. Primary Outcome: Elimination Half-life (t1/2) of Tazobactam
Description: Blood was collected for the determination of t1/2 of tazobactam. t1/2 is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 1 | 5 | 5 | 1 | 3
Hours | 0.702 (38.7) | 0.544 (3.1) | 0.719 (29.7) | 0.770 (34.2) | 0.538 (NA) — Cannot be calculated for n=1 | 0.815 (85.1) | 1.09 (32.0) | 3.03 (NA) — Cannot be calculated for n=1 | 0.875 (20.4)

15. Primary Outcome: Volume of Distribution at Steady State (Vss) of Ceftolozane
Description: Blood was collected for the determination of Vss of ceftolozane. Vss is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
L/kg | 0.274 (25.7) | 0.296 (22.0) | 0.331 (15.6) | 0.312 (19.5) | 0.282 (NA) — Cannot be calculated for n=1 | 0.340 (21.1) | 0.394 (12.6) | 0.344 (36.6) | 0.388 (26.9)

16. Primary Outcome: Volume of Distribution at Steady State (Vss) of Tazobactam
Description: Blood was collected for the determination of Vss of tazobactam. Vss is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 1 | 5 | 5 | 1 | 3
L/kg | 0.474 (69.6) | 0.740 (30.2) | 0.488 (32.0) | 0.513 (49.2) | 0.421 (NA) — Cannot be calculated for n=1 | 0.574 (36.2) | 0.668 (19.8) | 0.338 (NA) — Cannot be calculated for n=1 | 0.667 (29.3)

17. Primary Outcome: Plasma Clearance (CL) of Ceftolozane
Description: Blood was collected for the determination of CL of ceftolozane. CL is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour/kg
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 6 | 3 | 3 | 1 | 5 | 6 | 2 | 3
L/hour/kg | 0.146 (27.0) | 0.168 (21.3) | 0.181 (3.8) | 0.162 (31.1) | 0.176 (NA) — Cannot be calculated for n=1 | 0.149 (43.2) | 0.118 (36.0) | 0.0723 (32.2) | 0.147 (6.8)

18. Primary Outcome: Plasma Clearance (CL) of Tazobactam
Description: Blood was collected for the determination of CL of tazobactam. CL is expressed as geometric mean and percent geometric coefficient of variation, CV% = 100*sqrt(exp(s^2)-1), where s^2 is the observed between-subjects variance on the natural log-scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour/kg
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 1 | 5 | 5 | 1 | 3
L/hour/kg | 0.556 (53.9) | 0.886 (23.1) | 0.506 (42.0) | 0.519 (44.8) | 0.611 (NA) — Cannot be calculated for n=1 | 0.502 (34.7) | 0.385 (34.1) | 0.0760 (NA) — Cannot be calculated for n=1 | 0.452 (24.9)

19. Secondary Outcome: Number of Participants With One or More Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to Day 10
Population: The safety population was all enrolled participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 6 | 6 | 3 | 3 | 1 | 5 | 7 | 2 | 4
Participants | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 0

20. Secondary Outcome: Number of Participants Who Discontinued the Study Due to an Adverse Event
Description: as for outcome 19
Time Frame: Up to Day 10
Population: The safety population was all enrolled participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
Number analyzed (Participants) | 6 | 6 | 3 | 3 | 1 | 5 | 7 | 2 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 10
Description: The safety population was all enrolled participants who received study drug.
Arm/Group | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/3 | 0/3 | 0/1 | 0/5 | 0/7 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 0/3 | 0/3 | 0/1 | 1/5 | 0/7 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 1/3 | 1/3 | 1/1 | 1/5 | 1/7 | 2/2 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC (N=6) | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg (N=6) | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg (N=3) | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg (N=3) | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg (N=1) | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg (N=5) | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg (N=7) | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg (N=2) | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg (N=4)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ≥12 to <18 Years TOL/TAZ 1000/500 mg FDC (N=6) | Cohort 2: ≥7 to <12 Years TOL/TAZ 18/9 mg/kg (N=6) | Cohort 3: ≥2 to <7 Years TOL/TAZ 18/9 mg/kg (N=3) | Cohort 3: ≥2 to <7 Years TOL/TAZ 30/15 mg/kg (N=3) | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 18/9 mg/kg (N=1) | Cohort 4: ≥3 Months to <2 Years TOL/TAZ 30/15 mg/kg (N=5) | Cohort 5: Birth to <3 Months TOL/TAZ 20/10 mg/kg (N=7) | Cohort 6: Birth to <3 Months TOL/TAZ 12/6 mg/kg (N=2) | Cohort 6: Birth to <3 Months TOL/TAZ 20/10 mg/kg (N=4)
Waist circumference increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weaning failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device leakage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the Sponsor and are confidential. The Sponsor will make all reasonable efforts to publish the results of the study in an appropriate peer-reviewed journal. Authorship on the primary publication of the results from this study will be based on contributions to study design, enrollment, data analysis, and interpretation of results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02266706/Prot_SAP_000.pdf